CLINICAL TRIAL: NCT00523692
Title: Remission Induction in Very Early Rheumatoid Arthritis: a Comparison of Etanercept Plus Methotrexate Plus Steroid With Standard Therapy
Brief Title: Remission Induction in Very Early Rheumatoid Arthritis
Acronym: RIVERA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRK2939; REC reference 06/Q2404/95; EudraCT number 2006-001428-38; CTA number 16719/0201/001-0001
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Early arthritis; Rheumatoid arthritis; Rheumatoid factor; Anti CCP antibody; Remission; Anti-TNF therapy; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intensive therapy
  Interventions: Drug: Etanercept, methotrexate and depomedrone
- 2 (Active Comparator): Standard therapy
  Interventions: Drug: depemedrone

INTERVENTIONS:
Drug: Etanercept, methotrexate and depomedrone — Etanercept (50mg weekly; subcutaneous) Methotrexate (7.5-25mg weekly; oral) Depomedrone (up to 120mg; intraarticular / intramuscular)
  Arms: 1
Drug: depemedrone — depomedrone (up to 120mg im/ia) methotrexate (added after symptoms have been present for 12 weeks)
  Arms: 2

SUMMARY:
Rheumatoid arthritis (RA) is a debilitating chronic immune mediated inflammatory disease which affects 1% of the European population. RA is associated with significant joint damage, disability and an enhanced mortality. Current treatment strategies target patients once synovitis has been present for several months and it is clear that the patient has developed persistent disease. After the first 3 months of symptoms, we and others have shown that the persistence of chronic inflammation in the rheumatoid synovium is driven by hyperplastic stromal tissue which inhibits leukocyte apoptosis leading to the accumulation of inflammatory cells in the joint. Therapies at this stage of disease, with conventional disease modifying anti-rheumatic drugs (DMARDs) as well as drugs targeting TNF-alpha reduce disease activity but are unable to cure RA. We have now identified that the very early phase of synovitis in patients destined to develop RA (within the first 12 weeks of symptoms) represents a pathologically distinct phase of disease. This suggests that late disease is not just more of early disease and gives, for the first time, a clear rationale for very early intervention. Building on these recent observations, we propose to test the hypothesis that the disease processes in the very early stages of RA are fundamentally different to those in established chronic disease. This will be done by assessing whether treatment during this phase with the well-established gold standard modality of anti-TNF-alpha therapy and methotrexate can permanently switch off inflammation, preventing the development of RA and thereby effecting a cure of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Synovial swelling of at least 1 joint confirmed by clinical assessment
* Duration of symptoms attributable to inflammatory joint disease (pain, swelling or early morning stiffness of >1 hour) of < 12 weeks.
* Seropositivity for RF and anti-CCP Ab
* Women of childbearing potential or men capable of fathering children must be using adequate birth control measures (eg, abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, surgical sterilization) during the study.
* Female subjects of childbearing potential must test negative for pregnancy

Exclusion Criteria:

* Previous history of inflammatory arthritis.
* Previous use of DMARDs or anti-TNF-agents.
* Any current inflammatory condition with signs or symptoms that might confound the diagnosis (e.g. connective tissue disorders).
* Clinical evidence of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, prior to study entry.
* Administration, or expected administration, of any live virus or bacterial vaccination within 3 months before the first administration of study agent, or during the trial.
* A history of an infected joint prosthesis, or administration of antibiotics for a suspected infection of a joint prosthesis, if that prosthesis has not been removed or replaced.
* Known infection with HIV, hepatitis B, or hepatitis C.
* A serious infection that in the opinion of the investigator precludes receipt of a TNF blocking agent.
* Serious and uncontrolled co-existing disease that in the opinion of the investigator preclude the use of TNF-blocking medication, methotrexate or depomedrone (including pulmonary disease on chest radiograph, congestive cardiac failure (NYHA grade 3 or 4), history of demyelinating disease such as multiple sclerosis or optic neuritis).
* Bleeding disorder of the use of anti-coagulants
* Any known malignancy or a history of malignancy within the previous 5 years (with the exception of a basal cell carcinoma that has been treated with no evidence of recurrence).
* Any other contraindication to etanercept, methotrexate or parenteral depomedrone.
* Patients will also be excluded with the following laboratory results: haemoglobin <8.5 gm/dl, total white cell count <3.5 x 109/litre, serum transaminase value more than twice the upper limit of normal, and serum creatinine >150 micromoles/litre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-09

PRIMARY OUTCOMES:
The percentage of patients in drug free clinical remission at week 48 having withdrawn therapy at week 24 i.e. the induction of drug free remission. | week 48

SECONDARY OUTCOMES:
The percentage of patients in clinical remission at week 24 (when all drugs will be withdrawn if remission has been achieved). | week 24
The percentage of patients in radiological remission (no ultrasound evidence of synovitis) at week 24. | week 24
Clinical disease activity measures, including ACR responder rates (20%, 50%, and 70%), Disease Activity Score in 28 joints (DAS28), functional assessments (HAQ) and health status (EuroQuol-5D) at week 24. | week 24
The percentage of patients in drug free radiological remission (no ultrasound evidence of synovitis) at week 48 having withdrawn therapy at week 24. | week 48
Clinical disease activity measures, including ACR responder rates (20%, 50%, and 70%), Disease Activity Score in 28 joints (DAS28), functional assessments (HAQ) and health status (EuroQuol-5D) at weeks 48 and 96. | weeks 48 and 96.
The rate of progression of radiological change on conventional radiographs from baseline to week 48 and week 96. | weeks 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Karim Raza, MRCP PhD, Principal Investigator — University of Birmingham; Christopher D Buckley, FRCP PhD, Study Director — University of Birmingham
Locations (2):
- United Kingdom (2):
  - University Hopsital Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Sandwell and West Birmingham Hospitals NHS Trust, Birmingham, West Midlands

REFERENCES:
- [Background] Raza K, Falciani F, Curnow SJ, Ross EJ, Lee CY, Akbar AN, Lord JM, Gordon C, Buckley CD, Salmon M. Early rheumatoid arthritis is characterized by a distinct and transient synovial fluid cytokine profile of T cell and stromal cell origin. Arthritis Res Ther. 2005;7(4):R784-95. doi: 10.1186/ar1733. Epub 2005 Apr 7. PMID 15987480
- [Background] Raza K, Breese M, Nightingale P, Kumar K, Potter T, Carruthers DM, Situnayake D, Gordon C, Buckley CD, Salmon M, Kitas GD. Predictive value of antibodies to cyclic citrullinated peptide in patients with very early inflammatory arthritis. J Rheumatol. 2005 Feb;32(2):231-8. PMID 15693082
- [Background] Raza K, Buckley CE, Salmon M, Buckley CD. Treating very early rheumatoid arthritis. Best Pract Res Clin Rheumatol. 2006 Oct;20(5):849-63. doi: 10.1016/j.berh.2006.05.005. PMID 16980210